CLINICAL TRIAL: NCT05435339
Title: First-in-Human, Open-label, Dose-Escalation Trial With an Expansion Cohort to Evaluate the Safety of GEN1053 as Monotherapy in Subjects With Malignant Solid Tumors
Brief Title: A Study to Evaluate Safety, Tolerability, and Preliminary Effect of the GEN1053 Antibody on Malignant Solid Tumors as Monotherapy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to strategic evaluation of GEN1053 within the context of Genmab's portfolio
Sponsor: Genmab (Industry)
Collaborators: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCT1053-01; 2021-006692-42 (EudraCT Number); 1005700 (Other: IRAS ID; UK Research Summaries Database); 2022-502419-12-00 (EU CTIS Number)
Record Dates: First submitted 2022-06-23; First posted 2022-06-28 (Actual); Results first posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumor, Adult
Keywords: Monoclonal antibody

STUDY DESIGN:
Intervention Model Description: Sequential assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GEN1053 Monotherapy (Experimental)
  Interventions: Biological: GEN1053

INTERVENTIONS:
Biological: GEN1053 — GEN1053 will be administered as an intravenous (IV) infusion every 3rd week. The dose levels will be determined by the starting dose and the escalation steps taken in the trial.

SUMMARY:
The drug that will be investigated in the study is GEN1053. GEN1053 is an antibody designed to (re)activate and increase antitumor immunity.

Since this is the first study of GEN1053 in humans, the main purpose is to evaluate safety. Besides safety, the study will determine the recommended GEN1053 dose to be tested in a larger group of participants and assess preliminary clinical activity of GEN1053.

GEN1053 will be studied in a broad group of cancer patients, having different kinds of solid tumors. All participants will get GEN1053. The study consists of two parts: Part 1 tests increasing doses of GEN1053 ("escalation"), followed by Part 2 which tests the recommended phase 2 dose GEN1053 dose from Part 1 ("expansion").

DETAILED DESCRIPTION:
The trial is a First in Human open-label, multicenter, multinational safety trial in participants with non-central nervous system (non-CNS) metastatic or advanced malignant solid tumors for whom there is no available standard therapy likely to confer clinical benefit, evaluating the safety, tolerability, preliminary antitumor activity, pharmacokinetics (PK), pharmacodynamics (PD), and immunogenicity of GEN1053.

The trial will be conducted as follows:

* The Dose Escalation part (Part 1) will explore the safety of escalating doses of GEN1053 as monotherapy (phase 1)
* The Expansion part (Part 2) is planned to provide additional safety and initial antitumor activity information of the Recommended Phase 2 dose (RP2D) for GEN1053 monotherapy in selected tumor indications, as well as more detailed data related to the mode of action (MoA).

ELIGIBILITY:
Key Inclusion Criteria:

For both the Dose Escalation and Expansion parts:

* Be ≥18 years of age.
* Have measurable disease according to RECIST 1.1
* Provide all pre-baseline scans since failure of last prior therapy (ie radiographic PD), if available
* Have Eastern Cooperative Oncology Group performance status ≤1.
* Have organ and bone marrow function as follows:

Bone marrow / hematological function:

* Absolute neutrophil count (ANC) ≥1.5×10^9/L
* Hemoglobin ≥9.0 g/dL
* Platelet count ≥150×10^9/L

Liver function:

* Total bilirubin ≤ upper limit of normal (ULN)
* Alanine aminotransferase ≤1.5×ULN
* Aspartate aminotransferase ≤1.5×ULN
* Albumin ≥30 g/L

Coagulation status:

* Prothrombin time (PT)/International normalized ratio ≤1.5
* Activated partial thromboplastin time (aPTT) ≤1.5×ULN
* Renal function: Glomerular filtration rate ≥45 mL/min/1.73 m², according to the abbreviated Modification of Diet in Renal Disease equation

For Monotherapy Dose Escalation (phase 1) only:

* Subjects with histologically or cytologically confirmed non-CNS solid tumors that are metastatic or advanced.
* Subjects who have progressed on standard of care therapy or for whom there is no available standard therapy likely to provide clinical benefit, or who are not candidates for or refuse such available therapy, and for whom, in the opinion of the investigator, experimental therapy with GEN1053 may be beneficial.
* Fresh biopsies mandatory for all patients in Monotherapy Dose Escalation

For the Expansion part Only:

•Subjects with histologically or cytologically confirmed diagnosis of recurrent, unresectable or metastatic HNSCC, who have progressed on standard of care therapy or do not have any further available standard therapy or are not candidates for or refuse standard therapy (if subjects had access), and for whom experimental therapy with GEN1053 may be beneficial in the opinion of the investigator.

Key Exclusion Criteria (all parts):

* Has uncontrolled intercurrent illness, including but not limited to:

  * Ongoing or active infection requiring IV treatment with anti-infective therapy administered less than 2 weeks prior to first dose.
  * Symptomatic congestive heart failure (Grade III or IV as classified by the New York Heart Association), unstable angina pectoris or cardiac arrhythmia.
  * Uncontrolled hypertension defined as systolic blood pressure ≥160 mm Hg and/or diastolic blood pressure ≥100 mm Hg, despite optimal medical management.
  * Prolonged QTc interval at baseline of ≥470 milliseconds using Fridericia's QT correction formula.
  * Ongoing or recent (within 1 year) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments, which may suggest risk for irAEs.
  * History of grade 3 or higher irAEs that led to treatment discontinuation of a CPI.
  * History of chronic liver disease or evidence of hepatic cirrhosis.
  * Evidence of interstitial lung disease.
  * Ongoing pneumonitis or history of non-infectious pneumonitis that has required steroids.
  * Known platelet function defects
* Prior therapy:

  * Radiotherapy within 14 days prior to first GEN1053 administration. Palliative radiotherapy will be allowed.
  * Treatment with an anti-cancer agent (within 28 days or after at least 5 half-lives of the drug, whichever is shorter), prior to GEN1053 administration.
  * Subject with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of first treatment. Inhaled or topical steroids, and adrenal or pituitary replacement steroid > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - Yale University, New Haven, Connecticut
  - Sarah Cannon Research Institute, Nashville, Tennessee
- Spain (3):
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Centro Integral Oncologico Clara Campal, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results Summary in Plain Language — https://euclinicaltrials.eu/search-for-clinical-trials/?lang=en&EUCT=2022-502419-12-00

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was early terminated and only the GEN1053 monotherapy dose escalation was initiated and completed. The study was terminated prior to the start of the Dose Expansion Phase.
Groups:
- GEN1053 Dose Level 1 Once Every 3 Weeks (Q3W): Participants with malignant solid tumors were treated with dose level 1 of GEN1053 Q3W by intravenous (IV) infusion. Dose Level 1 was the lowest dose, and doses were increased incrementally up to Dose Level 8, which was the highest dose.
- GEN1053 Dose Level 2 Q3W: Participants with malignant solid tumors were treated with dose level 2 of GEN1053 Q3W by IV infusion. Dose Level 1 was the lowest dose, and doses were increased incrementally up to Dose Level 8, which was the highest dose.
- GEN1053 Dose Level 3 Q3W: Participants with malignant solid tumors were treated with dose level 3 of GEN1053 Q3W by IV infusion. Dose Level 1 was the lowest dose, and doses were increased incrementally up to Dose Level 8, which was the highest dose.
- GEN1053 Dose Level 4 Q3W: Participants with malignant solid tumors were treated with dose level 4 of GEN1053 Q3W by IV infusion. Dose Level 1 was the lowest dose, and doses were increased incrementally up to Dose Level 8, which was the highest dose.
- GEN1053 Dose Level 5 Q3W: Participants with malignant solid tumors were treated with dose level 5 of GEN1053 Q3W by IV infusion. Dose Level 1 was the lowest dose, and doses were increased incrementally up to Dose Level 8, which was the highest dose.
- GEN1053 Dose Level 6 Q3W: Participants with malignant solid tumors were treated with dose level 6 of GEN1053 Q3W by IV infusion. Dose Level 1 was the lowest dose, and doses were increased incrementally up to Dose Level 8, which was the highest dose.
- GEN1053 Dose Level 7 Q3W: Participants with malignant solid tumors were treated with dose level 7 of GEN1053 Q3W by IV infusion. Dose Level 1 was the lowest dose, and doses were increased incrementally up to Dose Level 8, which was the highest dose.
- GEN1053 Dose Level 8 Q3W: Participants with malignant solid tumors were treated with dose level 8 of GEN1053 Q3W by IV infusion. Dose Level 1 was the lowest dose, and doses were increased incrementally up to Dose Level 8, which was the highest dose.
Period: Overall Study
Arm/Group | GEN1053 Dose Level 1 Once Every 3 Weeks (Q3W) | GEN1053 Dose Level 2 Q3W | GEN1053 Dose Level 3 Q3W | GEN1053 Dose Level 4 Q3W | GEN1053 Dose Level 5 Q3W | GEN1053 Dose Level 6 Q3W | GEN1053 Dose Level 7 Q3W | GEN1053 Dose Level 8 Q3W
Started | 1 | 1 | 3 | 1 | 6 | 3 | 7 | 9
Received at Least 1 Dose of Study Drug | 1 | 1 | 3 | 1 | 6 | 3 | 7 | 9
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 3 | 1 | 6 | 3 | 7 | 9
Not completed — Death | 1 | 0 | 3 | 1 | 3 | 2 | 4 | 6
Not completed — Sponsor Decision | 0 | 1 | 0 | 0 | 2 | 1 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Measured in the Full Analysis Set, which included all participants who received at least 1 dose of trial drug. Participants were analyzed according to the actual trial treatment received.
Groups:
- GEN1053 Dose Level 1 Q3W: Participants with malignant solid tumors were treated with dose level 1 of GEN1053 Q3W by IV infusion. Dose Level 1 was the lowest dose, and doses were increased incrementally up to Dose Level 8, which was the highest dose.
- Total: Total of all reporting groups
Arm/Group | GEN1053 Dose Level 1 Q3W | GEN1053 Dose Level 2 Q3W | GEN1053 Dose Level 3 Q3W | GEN1053 Dose Level 4 Q3W | GEN1053 Dose Level 5 Q3W | GEN1053 Dose Level 6 Q3W | GEN1053 Dose Level 7 Q3W | GEN1053 Dose Level 8 Q3W | Total
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 6 | 3 | 7 | 9 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 1 | 1 | 4 | 1 | 3 | 9 | 19
  >=65 years | 1 | 1 | 2 | 0 | 2 | 2 | 4 | 0 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 79 | 78 | 62.3 (13.9) | 57 | 55.2 (13.1) | 66 (16.1) | 68.7 (8.4) | 57 (5.7) | 62.1 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 0 | 4 | 2 | 5 | 4 | 16
  Male | 1 | 0 | 3 | 1 | 2 | 1 | 2 | 5 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Missing | 0 | 0 | 2 | 1 | 4 | 2 | 7 | 5 | 21
  Not Hispanic or Latino | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 4 | 8
  Not Reported | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 1 | 3 | 1 | 6 | 3 | 7 | 9 | 31
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 0 | 0 | 2 | 1 | 4 | 2 | 7 | 5 | 21
  United States of America (The) | 1 | 1 | 1 | 0 | 2 | 1 | 0 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: The occurrence of any of the following toxicities, assessed as related to trial treatment, were considered DLTs: All Grade 5 events, Grade 4 anaphylaxis, infusion-related reactions and neutropenia for ≥7 days, Grade 3/4 febrile neutropenia, Grade 4 thrombocytopenia, Grade 3 thrombocytopenia with clinically significant bleeding, Grade 4 anemia, Grade 4 aspartate aminotransferase (AST), alanine aminotransferase (ALT), or bilirubin elevation/Grade 3 that did not recover to ≤Grade 1 within 14 days, AST or ALT elevations ≥Grade 2 with concomitant bilirubin >2.0×upper limit of normal with no signs of cholestasis, any Grade 4 immune-related adverse event (irAE), Grade 3 irAEs that did not improve to ≤Grade 1 within 7 days (with exceptions), Grade 4 cytokine release syndrome (CRS), Grade 3 CRS not resolved to ≤Grade 2 within 48 hrs following adequate intervention, any other ≥Grade 3 nonhematological adverse event (AE) during the first GEN1053 treatment cycle (with exceptions), cycle=3 weeks.
Time Frame: Day 1 up to Day 21
Population: Measured in the Safety Analysis Set, which included all participants who received at least 1 dose of trial drug. Participants were analyzed according to the actual trial treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | GEN1053 Dose Level 1 Q3W | GEN1053 Dose Level 2 Q3W | GEN1053 Dose Level 3 Q3W | GEN1053 Dose Level 4 Q3W | GEN1053 Dose Level 5 Q3W | GEN1053 Dose Level 6 Q3W | GEN1053 Dose Level 7 Q3W | GEN1053 Dose Level 8 Q3W
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 6 | 3 | 7 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

2. Primary Outcome: Number of Participants With At Least One Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical trial participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE was therefore any unfavorable and unintended sign (including an abnormal safety laboratory parameter finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. A TEAE was defined as an AE occurring or worsening after first dose. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to approximately 1.5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GEN1053 Dose Level 1 Q3W | GEN1053 Dose Level 2 Q3W | GEN1053 Dose Level 3 Q3W | GEN1053 Dose Level 4 Q3W | GEN1053 Dose Level 5 Q3W | GEN1053 Dose Level 6 Q3W | GEN1053 Dose Level 7 Q3W | GEN1053 Dose Level 8 Q3W
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 6 | 3 | 7 | 9
Participants | 1 | 1 | 3 | 1 | 6 | 3 | 7 | 9

3. Secondary Outcome: Clearance (CL) of GEN1053
Description: Venous blood samples were collected for analyzing the pharmacokinetics (PK) of GEN1053.
Time Frame: Cycle 1 and Cycle 3 (cycles were 3 weeks)
Population: Measured in the Pharmacokinetic (PK) Analysis Set, which included all participants who received at least 1 dose of trial drug and who provided at least 1 evaluable PK sample. Overall number of participants analyzed = participants with evaluable data for the outcome measure. Number analyzed = participants with evaluable data at the specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliters (mL)/day
Arm/Group | GEN1053 Dose Level 1 Q3W | GEN1053 Dose Level 2 Q3W | GEN1053 Dose Level 3 Q3W | GEN1053 Dose Level 4 Q3W | GEN1053 Dose Level 5 Q3W | GEN1053 Dose Level 6 Q3W | GEN1053 Dose Level 7 Q3W | GEN1053 Dose Level 8 Q3W
Number analyzed (Participants) | 1 | 1 | 3 | 0 | 6 | 3 | 7 | 9
milliliters (mL)/day
  Cycle 1 | 2450.0 | 3120.0 | 916.7 (30.8) |  | 594.0 (19.7) | 491.3 (35.6) | 471.7 (29.5) | 567.7 (39.1)
  Cycle 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 2
  Cycle 3 |  |  |  |  | 293.1 (19.5) |  | 244.5 (36.0) | 435.2 (27.3)

4. Secondary Outcome: Volume of Distribution (Vz) of GEN1053
Description: Venous blood samples were collected for analyzing concentrations of GEN1053.
Time Frame: Cycle 1 and Cycle 3 (cycles were 3 weeks)
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL
Arm/Group | GEN1053 Dose Level 1 Q3W | GEN1053 Dose Level 2 Q3W | GEN1053 Dose Level 3 Q3W | GEN1053 Dose Level 4 Q3W | GEN1053 Dose Level 5 Q3W | GEN1053 Dose Level 6 Q3W | GEN1053 Dose Level 7 Q3W | GEN1053 Dose Level 8 Q3W
Number analyzed (Participants) | 1 | 1 | 3 | 0 | 6 | 3 | 7 | 9
mL
  Cycle 1 | 4300.0 | 3950.0 | 6077.1 (17.9) |  | 6108.9 (34.2) | 6455.8 (8.1) | 6808.7 (73.4) | 7434.6 (70.8)
  Cycle 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 2
  Cycle 3 |  |  |  |  | 5683.6 (36.1) |  | 5302.1 (9.1) | 10834.8 (77.5)

5. Secondary Outcome: Maximum (Peak) Concentration (Cmax) of GEN1053
Description: Venous blood samples were collected for analyzing concentrations of GEN1053.
Time Frame: Cycle 1 and Cycle 3 (cycles were 3 weeks)
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms (μg)/mL
Arm/Group | GEN1053 Dose Level 1 Q3W | GEN1053 Dose Level 2 Q3W | GEN1053 Dose Level 3 Q3W | GEN1053 Dose Level 4 Q3W | GEN1053 Dose Level 5 Q3W | GEN1053 Dose Level 6 Q3W | GEN1053 Dose Level 7 Q3W | GEN1053 Dose Level 8 Q3W
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 6 | 3 | 7 | 9
micrograms (μg)/mL
  Cycle 1 | 0.530 | 1.570 | 5.583 (27.187) | 12.000 | 16.862 (8.824) | 60.854 (44.313) | 124.869 (22.050) | 218.641 (24.465)
  Cycle 3: number analyzed (Participants) | 0 | 1 | 0 | 0 | 3 | 1 | 3 | 3
  Cycle 3 |  | 1.450 |  |  | 20.970 (11.732) | 60.400 | 159.509 (26.510) | 306.525 (31.455)

6. Secondary Outcome: Time to Maximum (Peak) Concentration (Tmax) of GEN1053
Description: Venous blood samples were collected for analyzing concentrations of GEN1053.
Time Frame: Cycle 1 and Cycle 3 (cycles were 3 weeks)
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | GEN1053 Dose Level 1 Q3W | GEN1053 Dose Level 2 Q3W | GEN1053 Dose Level 3 Q3W | GEN1053 Dose Level 4 Q3W | GEN1053 Dose Level 5 Q3W | GEN1053 Dose Level 6 Q3W | GEN1053 Dose Level 7 Q3W | GEN1053 Dose Level 8 Q3W
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 6 | 3 | 7 | 9
days
  Cycle 1 | 0.0620 | 0.0600 | 0.0583 (3.5988) | 0.1390 | 0.0855 (65.5230) | 0.0760 (45.9942) | 0.0826 (75.6636) | 0.0953 (60.7249)
  Cycle 3: number analyzed (Participants) | 0 | 1 | 0 | 0 | 3 | 1 | 3 | 3
  Cycle 3 |  | 0.1350 |  |  | 0.1023 (64.0898) | 0.1390 | 0.0784 (43.4302) | 0.0746 (49.4225)

7. Secondary Outcome: Predose Trough Concentration (Ctrough) of GEN1053
Description: Venous blood samples were collected for analyzing concentrations of GEN1053.
Time Frame: Cycle 1 and Cycle 3 (cycles were 3 weeks)
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | GEN1053 Dose Level 1 Q3W | GEN1053 Dose Level 2 Q3W | GEN1053 Dose Level 3 Q3W | GEN1053 Dose Level 4 Q3W | GEN1053 Dose Level 5 Q3W | GEN1053 Dose Level 6 Q3W | GEN1053 Dose Level 7 Q3W | GEN1053 Dose Level 8 Q3W
Number analyzed (Participants) | 1 | 1 | 3 | 0 | 5 | 2 | 3 | 5
ug/mL
  Cycle 1 | 0.0250 | 0.0250 | 0.1322 (58.7685) |  | 1.5722 (60.7405) | 6.0890 (132.2920) | 24.8853 (4.2283) | 33.6922 (28.1602)
  Cycle 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 1
  Cycle 3 |  |  |  |  | 4.3705 (53.5677) |  | 58.5326 (12.2317) | 56.3000

8. Secondary Outcome: Elimination Half-life (t1/2) of GEN1053
Description: Venous blood samples were collected for analyzing concentrations of GEN1053.
Time Frame: Cycle 1 and Cycle 3 (cycles were 3 weeks)
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | GEN1053 Dose Level 1 Q3W | GEN1053 Dose Level 2 Q3W | GEN1053 Dose Level 3 Q3W | GEN1053 Dose Level 4 Q3W | GEN1053 Dose Level 5 Q3W | GEN1053 Dose Level 6 Q3W | GEN1053 Dose Level 7 Q3W | GEN1053 Dose Level 8 Q3W
Number analyzed (Participants) | 1 | 1 | 3 | 0 | 6 | 3 | 7 | 9
days
  Cycle 1 | 1.2200 | 0.8750 | 4.5977 (13.0224) |  | 7.1235 (53.5614) | 9.1195 (30.0207) | 10.0111 (81.6893) | 9.0787 (100.0112)
  Cycle 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 2
  Cycle 3 |  |  |  |  | 13.4236 (53.5705) |  | 15.0597 (27.0838) | 17.2624 (43.0077)

9. Secondary Outcome: Area Under the Concentration-time Curve (AUC) From Time Zero to Last Quantifiable Measurement (AUClast) of GEN1053
Description: Venous blood samples were collected for analyzing concentrations of GEN1053.
Time Frame: Cycle 1 and Cycle 3 (cycles were 3 weeks)
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/mL
Arm/Group | GEN1053 Dose Level 1 Q3W | GEN1053 Dose Level 2 Q3W | GEN1053 Dose Level 3 Q3W | GEN1053 Dose Level 4 Q3W | GEN1053 Dose Level 5 Q3W | GEN1053 Dose Level 6 Q3W | GEN1053 Dose Level 7 Q3W | GEN1053 Dose Level 8 Q3W
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 6 | 3 | 7 | 9
day*ug/mL
  Cycle 1 | 0.5620 | 1.5300 | 21.8315 (30.8860) | 15.2000 | 86.0185 (62.0662) | 379.6819 (41.9278) | 678.2510 (55.6633) | 1190.8115 (69.3078)
  Cycle 3: number analyzed (Participants) | 0 | 1 | 0 | 0 | 3 | 1 | 3 | 3
  Cycle 3 |  | 0.1930 |  |  | 204.3491 (19.5536) | 423.0000 | 1510.1353 (51.8536) | 1985.3056 (33.6209)

10. Secondary Outcome: AUC From Time Zero Over the Dosing Interval (AUCtau) of GEN1053
Description: Venous blood samples were collected for analyzing concentrations of GEN1053.
Time Frame: Cycle 1 and Cycle 3 (cycles were 3 weeks)
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/mL
Arm/Group | GEN1053 Dose Level 1 Q3W | GEN1053 Dose Level 2 Q3W | GEN1053 Dose Level 3 Q3W | GEN1053 Dose Level 4 Q3W | GEN1053 Dose Level 5 Q3W | GEN1053 Dose Level 6 Q3W | GEN1053 Dose Level 7 Q3W | GEN1053 Dose Level 8 Q3W
Number analyzed (Participants) | 1 | 1 | 3 | 0 | 6 | 3 | 7 | 9
day*ug/mL
  Cycle 1 | 0.8170 | 1.9200 | 21.8315 (30.8860) |  | 100.5407 (19.7816) | 402.5411 (37.4881) | 835.4647 (28.4628) | 1392.1084 (37.2599)
  Cycle 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 2
  Cycle 3 |  |  |  |  | 203.9020 (19.9691) |  | 1656.9616 (36.6222) | 1842.9867 (26.7838)

11. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADAs) to GEN1053
Description: Venous blood samples were drawn for analysis of ADAs in serum samples.
Time Frame: Cycle 1 Day 1 through end of safety follow up (60 days after last dose [cycles were 3 weeks]), up to approximately 1.5 years
Population: Measured in the Pharmacokinetic (PK) Analysis Set, which included all participants who received at least 1 dose of trial drug and who provided at least 1 evaluable PK sample. Overall number of participants analyzed = participants with evaluable data for the outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | GEN1053 Dose Level 1 Q3W | GEN1053 Dose Level 2 Q3W | GEN1053 Dose Level 3 Q3W | GEN1053 Dose Level 4 Q3W | GEN1053 Dose Level 5 Q3W | GEN1053 Dose Level 6 Q3W | GEN1053 Dose Level 7 Q3W | GEN1053 Dose Level 8 Q3W
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 6 | 3 | 7 | 9
Participants
  Cycle 1 Day 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 3 Day 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 4 Day 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 6 Day 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 8 Day 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 10 Day 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 12 Day 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 14 Day 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 16 Day 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 18 Day 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 20 Day 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  End of Treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Safety Follow Up 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Safety Follow Up 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the number of participants with best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR) (ie, "responders"), as per local review and according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR was defined as all of the following: disappearance of all target and non-target tumor lesions, and reduction in short axis to <10 millimeters (mm) in all pathological target and non-target lymph nodes, and normalization of tumor marker level (if applicable). PR was defined as ≥30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Data are presented for the number of participants with ORR.
Time Frame: Up to approximately 1.5 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | GEN1053 Dose Level 1 Q3W | GEN1053 Dose Level 2 Q3W | GEN1053 Dose Level 3 Q3W | GEN1053 Dose Level 4 Q3W | GEN1053 Dose Level 5 Q3W | GEN1053 Dose Level 6 Q3W | GEN1053 Dose Level 7 Q3W | GEN1053 Dose Level 8 Q3W
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 6 | 3 | 7 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the number of participants with CR, PR, or stable disease (SD). CR was defined as all of the following: disappearance of all target and non-target tumor lesions, and reduction in short axis to <10 mm in all pathological target and non-target lymph nodes, and normalization of tumor marker level (if applicable). PR was defined as ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters (nadir) while on study. Data are presented for the number of participants with DCR.
Time Frame: Up to approximately 1.5 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | GEN1053 Dose Level 1 Q3W | GEN1053 Dose Level 2 Q3W | GEN1053 Dose Level 3 Q3W | GEN1053 Dose Level 4 Q3W | GEN1053 Dose Level 5 Q3W | GEN1053 Dose Level 6 Q3W | GEN1053 Dose Level 7 Q3W | GEN1053 Dose Level 8 Q3W
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 6 | 3 | 7 | 9
Participants | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 2

14. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the first documentation of objective tumor response (CR or PR) to the date of first PD or death due to any cause in participants whose confirmed BOR was CR or PR.
Time Frame: Up to approximately 1.5 years
Population: Measured in the Full Analysis Set (which included all participants who received at least 1 dose of trial drug) in those participants whose confirmed BOR was CR or PR. Participants were analyzed according to the actual trial treatment received. Overall number of participants analyzed = 0 as no participants had a confirmed BOR of CR or PR.
Arm/Group | GEN1053 Dose Level 1 Q3W | GEN1053 Dose Level 2 Q3W | GEN1053 Dose Level 3 Q3W | GEN1053 Dose Level 4 Q3W | GEN1053 Dose Level 5 Q3W | GEN1053 Dose Level 6 Q3W | GEN1053 Dose Level 7 Q3W | GEN1053 Dose Level 8 Q3W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 1.5 years
Description: Measured in the Safety Analysis Set, which included all participants who received at least 1 dose of trial drug. Participants were analyzed according to the actual trial treatment received.
Arm/Group | GEN1053 Dose Level 1 Q3W | GEN1053 Dose Level 2 Q3W | GEN1053 Dose Level 3 Q3W | GEN1053 Dose Level 4 Q3W | GEN1053 Dose Level 5 Q3W | GEN1053 Dose Level 6 Q3W | GEN1053 Dose Level 7 Q3W | GEN1053 Dose Level 8 Q3W
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/1 | 3/3 | 1/1 | 3/6 | 2/3 | 4/7 | 6/9
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/1 | 0/3 | 0/1 | 1/6 | 1/3 | 0/7 | 3/9
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 3/3 | 1/1 | 6/6 | 3/3 | 7/7 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GEN1053 Dose Level 1 Q3W (N=1) | GEN1053 Dose Level 2 Q3W (N=1) | GEN1053 Dose Level 3 Q3W (N=3) | GEN1053 Dose Level 4 Q3W (N=1) | GEN1053 Dose Level 5 Q3W (N=6) | GEN1053 Dose Level 6 Q3W (N=3) | GEN1053 Dose Level 7 Q3W (N=7) | GEN1053 Dose Level 8 Q3W (N=9)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune system disorder (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GEN1053 Dose Level 1 Q3W (N=1) | GEN1053 Dose Level 2 Q3W (N=1) | GEN1053 Dose Level 3 Q3W (N=3) | GEN1053 Dose Level 4 Q3W (N=1) | GEN1053 Dose Level 5 Q3W (N=6) | GEN1053 Dose Level 6 Q3W (N=3) | GEN1053 Dose Level 7 Q3W (N=7) | GEN1053 Dose Level 8 Q3W (N=9)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (6) | 1 (1) | 2 (3) | 4 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Face oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Blood fibrinogen decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (4) | 1 (2) | 4 (5) | 5 (19)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (3)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (4) | 4 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradyphrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 2 (2)
Abdominal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 1 (9)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procalcitonin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (2)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 2 (3) | 2 (7) | 2 (5) | 4 (15)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (5)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Klebsiella urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (15)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-07): https://cdn.clinicaltrials.gov/large-docs/39/NCT05435339/Prot_SAP_000.pdf